CLINICAL TRIAL: NCT02592473
Title: Prostate Artery Embolization Safety and Efficacy: A Pilot Study
Brief Title: Prostate Artery Embolization (PAE) for Treatment of Benign Prostatic Hyperplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Principal Investigator, Ziv Haskal, MD, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18236
Record Dates: First submitted 2015-10-26; First posted 2015-10-30 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Prostatic Hyperplasia; Benign Prostatic Hyperplasia (BPH); Prostatism; Lower Urinary Tract Symptoms (LUTS); Prostatic Hypertrophy; Hyperplasia; Male Urogenital Diseases; Genital Diseases, Male
Keywords: Prostate Artery Embolization (PAE); Benign Prostatic Hyperplasia (BPH); Lower Urinary Tract Symptoms (LUTS); BPH; PAE; LUTS; Prostatic Artery Embolization
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatism; Lower Urinary Tract Symptoms; Hyperplasia; Male Urogenital Diseases; Genital Diseases, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Embozene Microspheres (Experimental): Embozene Microspheres are spherical particles consisting of a hydrogel core and a poly nanocoat that will be used during study procedure, Prostatic Artery Embolization (PAE) to reduce or eliminate bloodflow to the prostate.
  Interventions: Device: Embozene Microspheres

INTERVENTIONS:
Device: Embozene Microspheres — Minimally invasive intra-arterial administration of particle embolics into prostate arteries under fluoroscopy and cone-beam CT imaging guidance.

SUMMARY:
The purpose of this project is to evaluate the safety, efficacy, and feasibility of performing prostatic artery embolization (PAE) using endovascular techniques and particle embolics in men suffering from lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
This pilot study is a prospective, non-randomized clinical trial assessing the safety and feasibility of prostatic artery embolization. Fifty adult male subjects will be enrolled and treated in this study. Patients who provide informed consent and are deemed eligible for participation will undergo prostatic artery embolization in the Interventional Radiology department at the University of Virginia. After performing an angiogram to identify the prostatic arteries, tiny particles known as Embozene Microspheres will be injected into the prostatic artery. Injecting these particles into the prostatic artery will slow blood flow to the prostate and thus shrinking the size of the prostate. By shrinking the size of the prostate, it is hopeful that it will provide relief of lower urinary tract symptoms due to BPH. Subjects will be followed for 2 years as part of their participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients between ages 45-80 years
* Diagnosis of Lower Urinary Tract Symptoms from Benign Prostatic Hypertrophy for a minimum of 6 months
* IPSS score at initial evaluation should be greater than 7, and uroflowmetry (Qmax) of <12mL/s (milliliters per second) .
* All prostate volumes will be at least 40gm and no more than 400gm based on DRE, TRUS, or cross sectional imaging

Exclusion Criteria:

* Patients with urinary tract infections (> 2/year), prostatitis, or interstitial cystitis
* Cases of biopsy proven prostate cancer or urethral cancer.
* Patients on long-term narcotic analgesia, androgen therapy, or GNRH (gonadotropin-releasing hormone) analogue therapy within 2 months of study.
* Patients who are classified as New York Heart Association Class III (Moderate), or higher.
* Patients with history of prior pelvic irradiation.
* Hypersensitivity reactions to contrast material not manageable with prophylaxis.
* Patients with serum creatinine values >1.7mg/dl or glomerular filtration rates less than 50.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement in Lower Urinary Tract Symptoms (LUTS) | 12 months
  QMax (peak urinary flow rate) assessment
Presence or absence of ischemic complications to the bladder, rectum, or other pelvic structures | 2 weeks
Clinical improvement in Lower Urinary Tract Symptoms (LUTS) | 24 months
  QMax assessment
Presence or absence of ischemic complications to the bladder, rectum, or other pelvic structures | 24 months
Clinical improvement in Lower Urinary Tract Symptoms (LUTS) | 12 months
  IPSS (International Prostate Symptom Score)
Clinical improvement in Lower Urinary Tract Symptoms (LUTS) | 24 months
  IPSS
Clinical improvement in Lower Urinary Tract Symptoms (LUTS) | 12 months
  QoL(quality of life question)
Clinical improvement in Lower Urinary Tract Symptoms (LUTS) | 24 months
  QoL
Clinical improvement in Lower Urinary Tract Symptoms (LUTS) | 24 months
  QMax

SECONDARY OUTCOMES:
Urine flow rate as measured by QMax | 1 month
Urine flow rate as measured by QMax | 24 months
Post-void residual measured in ml/cc | 1 month
Post-void residual measured in ml/cc | 24 months
UCLA-PCI-SF (University of California, Los Angeles Prostate Cancer Index Short Form) score | 1 month
UCLA-PCI-SF score | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ziv J Haskal, MD, Principal Investigator — Professor of Radiology
Locations (1):
- University of Virginia Health Systems, Charlottesville, Virginia, United States